CLINICAL TRIAL: NCT06149923
Title: Association Between ABO Polymorphism and Gastric/Colorectal Cancers
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Wesam Ashraf Soliman Ahmed, doctor, Assiut University
Other Study IDs: ABO in gastric/colorectal canc
Record Dates: First submitted 2023-11-19; First posted 2023-11-29 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Gastric Cancer; Colo-rectal Cancer
MeSH Terms: conditions — Stomach Neoplasms; Colonic Neoplasms | interventions — Real-Time Polymerase Chain Reaction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- cases: Patients that histopathologically confirmed gastric and/or colorectal cancer, males and females.
  Interventions: Genetic: quantitative Real-time PCR

INTERVENTIONS:
Genetic: quantitative Real-time PCR — : quantitative real time PCR using 7500 fast real time PCR (Applied Biosystems

SUMMARY:
To assess ABO gene polymorphism (rs8176746) in the patients histopathologically confirmed gastric and/or colorectal cancers relative to healthy controls by real time PCR.

DETAILED DESCRIPTION:
The ABO blood group system was discovered by the Austrian pathologist Karl Landsteiner in 1901, who classified the blood groups based on the presence of A and B antigens on the surface of red blood cells after noting patterns of agglutination during blood transfusion. Since the discovery of the ABO blood group system , several studies investigating the relationship between the ABO blood group system and various diseases have been conducted , cancer included .

First association between ABO blood group and cancer risk was reported in 1953 in The English patients with gastric cancer.

Gastric cancer is one of the most common malignant tumors of the digestive system , worldwide, gastric cancer is still the fourth most common cancer and the second most common cause of cancer death . The development of gastric cancer is caused by the interaction of genetic and environmental factors , ABO blood grouping is one of the most stable genetic factors.

This association is also observed with other gastrointestinal malignancies, including colorectal cancer which considered the third common cancer in both women and men and responsible for approximately 10% of all cancers, and the third most common cause of cancer related mortality for men and fourth for women .

The ABO is also the first blood group system defined at the gene level . SNP is a single nucleotide polymorphism, is a germ line substitution of a single nucleotide at a specific position in the genome that is present in a sufficiently large fraction of considered population , SNP may act as biological markers, as they can relate to the genes that are associated with various complex diseases as heart diseases, diabetes, cancer … etc.

In previous studies , significant association between ABO gene SNP (rs8176746) , H. Pylori infection, gastric and pancreatic cancer were found , as they observed that this gene SNP was associated with decreased risk of these disorders.

ELIGIBILITY:
Inclusion Criteria:

* Patients that histopathologically confirmed gastric and/or colorectal cancer.
* males and females.

Exclusion Criteria:

* Presence of other haematological , autoimmune disorders or other malignancies.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients that histopathologically confirmed gastric and/or colorectal cancer, males and females.
Sampling Method: Non-Probability Sample
Enrollment: 184 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
assess ABO gene polymorphism (rs8176746) in the patients histopathologically confirmed gastric and/colorectal cancers relative to healthy controls. | Baseline
  assess ABO gene polymorphism (rs8176746) in the patients histopathologically confirmed gastric and/colorectal cancers relative to healthy controls by real-time PCR.
  and determine the impact of ABO phenotype and genotype on risk of development of gastric and/or colorectal cancers.

REFERENCES:
- [Background] Groot HE, Villegas Sierra LE, Said MA, Lipsic E, Karper JC, van der Harst P. Genetically Determined ABO Blood Group and its Associations With Health and Disease. Arterioscler Thromb Vasc Biol. 2020 Mar;40(3):830-838. doi: 10.1161/ATVBAHA.119.313658. Epub 2020 Jan 23. PMID 31969017
- [Background] Rummel SK, Ellsworth RE. The role of the histoblood ABO group in cancer. Future Sci OA. 2016 Mar 15;2(2):FSO107. doi: 10.4155/fsoa-2015-0012. eCollection 2016 Jun. PMID 28031957
- [Background] Chen Z, Yang SH, Xu H, Li JJ. ABO blood group system and the coronary artery disease: an updated systematic review and meta-analysis. Sci Rep. 2016 Mar 18;6:23250. doi: 10.1038/srep23250. PMID 26988722
- [Background] Rummel S, Shriver CD, Ellsworth RE. Relationships between the ABO blood group SNP rs505922 and breast cancer phenotypes: a genotype-phenotype correlation study. BMC Med Genet. 2012 May 29;13:41. doi: 10.1186/1471-2350-13-41. PMID 22642827
- [Background] Zhou Y, Cui JG, Huang F, Zhang A, Li C, Zhao ZC, Li WD, Fu WH. Prognostic Factors for Survival in Node-Negative Gastric Cancer Patients Who Underwent Curative Resection. Scand J Surg. 2017 Sep;106(3):235-240. doi: 10.1177/1457496916677878. Epub 2017 Apr 4. PMID 28376652
- [Background] Crew KD, Neugut AI. Epidemiology of gastric cancer. World J Gastroenterol. 2006 Jan 21;12(3):354-62. doi: 10.3748/wjg.v12.i3.354. PMID 16489633
- [Background] Brenner H, Rothenbacher D, Arndt V. Epidemiology of stomach cancer. Methods Mol Biol. 2009;472:467-77. doi: 10.1007/978-1-60327-492-0_23. PMID 19107449
- [Background] Sano T, Coit DG, Kim HH, Roviello F, Kassab P, Wittekind C, Yamamoto Y, Ohashi Y. Proposal of a new stage grouping of gastric cancer for TNM classification: International Gastric Cancer Association staging project. Gastric Cancer. 2017 Mar;20(2):217-225. doi: 10.1007/s10120-016-0601-9. Epub 2016 Feb 20. PMID 26897166
- [Background] Urun Y, Ozdemir NY, Utkan G, Akbulut H, Savas B, Oksuzoglu B, Oztuna DG, Dogan I, Yalcin B, Senler FC, Onur H, Demirkazik A, Zengin N, Icli F. ABO and Rh blood groups and risk of colorectal adenocarcinoma. Asian Pac J Cancer Prev. 2012;13(12):6097-100. doi: 10.7314/apjcp.2012.13.12.6097. PMID 23464411
- [Background] Nakao M, Matsuo K, Ito H, Shitara K, Hosono S, Watanabe M, Ito S, Sawaki A, Iida S, Sato S, Yatabe Y, Yamao K, Ueda R, Tajima K, Hamajima N, Tanaka H. ABO genotype and the risk of gastric cancer, atrophic gastritis, and Helicobacter pylori infection. Cancer Epidemiol Biomarkers Prev. 2011 Aug;20(8):1665-72. doi: 10.1158/1055-9965.EPI-11-0213. Epub 2011 Jun 15. PMID 21680535
- [Background] Rizzato C, Campa D, Pezzilli R, Soucek P, Greenhalf W, Capurso G, Talar-Wojnarowska R, Heller A, Jamroziak K, Khaw KT, Key TJ, Bambi F, Landi S, Mohelnikova-Duchonova B, Vodickova L, Buchler MW, Bugert P, Vodicka P, Neoptolemos JP, Werner J, Hoheisel JD, Bauer AS, Giese N, Canzian F. ABO blood groups and pancreatic cancer risk and survival: results from the PANcreatic Disease ReseArch (PANDoRA) consortium. Oncol Rep. 2013 Apr;29(4):1637-44. doi: 10.3892/or.2013.2285. Epub 2013 Feb 12. PMID 23403949